CLINICAL TRIAL: NCT03750370
Title: Role of Colored Doppler Sonography in Evaluation of Testicular Perfusion Before and After Varicocelectomy in Patients With Infertility
Brief Title: Color Doppler in Varicocelectomy in Infertile Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammad Aly, Resident, Assiut University
Other Study IDs: doppler in varicocelectomy
Record Dates: First submitted 2018-11-18; First posted 2018-11-23 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Varicocelectomy; Doppler
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Doppler ultrasound — Colored Doppler Sonography is well established to illustrate microvascularity and therefore perfusion of the testis. The arterial flow velocities (peak systolic velocity [PSV] and end diastolic velocity [EDV]) and the resistance indices against this flow (resistive index [RI] and pulsatility index [PI]) in the testis can be measured with this technique.

SUMMARY:
To evaluate the long-term effects of varicocelectomy on testicular arterial flow via Color Doppler Sonography Parameters; The arterial flow velocities (peak systolic velocity [PSV] and end diastolic velocity [EDV]) and the resistance indices against this flow (resistive index [RI] and pulsatility index [PI]) of the testicular artery.

DETAILED DESCRIPTION:
Introduction Varicocele, an abnormal dilatation of the internal spermatic veins, is considered the major reversible cause of male infertility. It is observed in 35%-40% of all men with primary infertility and in up to 80% of those with secondary infertility.

The higher incidence of varicocele in men with secondary infertility suggests its progressive nature, which might be explained by a progressive testicular dysfunction involving both spermatogenesis and steroidogenesis. The negative impact of varicocele on spermatogenesis has been documented by a progressive reduction in the size of testicle ipsilateral to the varicocele.

Semen parameters improvement after varicocele treatment were first reported by Tulloch in the mid-20th century, who performed high surgical ligation of varicose veins in 30 patients with infertility. The author showed a marked improvement in postoperative seminal parameters in 66% of the treated subjects.

Several theories have been formulated to explain the testicular impairment caused by varicocele, including hypoxia, autoimmunity, elevated testicular temperature, reflux of catecholamine, and increased oxidative stress. However, none of them can completely explain the variable modulating effect of varicocele on male fertility. Recently, the oxidative stress theory has emerged as an important contributory factor due to findings of an association between elevated reactive oxygen species and impaired sperm function in men with varicocele. Additionally, reduction of oxidative stress markers has been noted after varicocele repair.

It is hypothesized that impaired venous drainage causes an increase in venous stasis and a decrease in arterial blood flow, thus inducing hypoxia and deficiency in testicular microcirculation . Also, it is thought that this hypoxia could be responsible for defective energy metabolism at mitochondrial levels, causing dysfunction of both Leydig and germinal cells.

The arterial supply to the human testis has 3 major components: the testicular artery, the cremasteric artery, and the vasal artery. Two-thirds of total blood is supplied by the testicular artery. The testicular artery divides into 2 branches in the testis; the capsular branch continues in the surface of the testis, the intratesticular branch continues in the parenchyma and deep into the testis.

Colored Doppler Sonography is well established to illustrate microvascularity and therefore perfusion of the testis. The arterial flow velocities (peak systolic velocity [PSV] and end diastolic velocity [EDV]) and the resistance indices against this flow (resistive index [RI] and pulsatility index [PI]) in the testis can be measured with this technique.

The encouraging benefits of varicocele repair to the semen parameters of subfertile men were ratified by three recent meta-analyses:

Agarwal et al. pooled 17 studies that included only infertile men with clinical varicocele and with at least one abnormal semen parameter. The intervention was either high ligation of the veins or subinguinal microsurgical varicocelectomy. There was a consistent improvement in sperm concentration and motility after both high ligation and microsurgical subinguinal techniques, with better results after microsurgical approach. Sperm morphology change was not stratified according to the type of intervention; nevertheless, there was an increment of 3.16% on the average of normal forms.

Baazeem et al. have also evaluated the role of varicocele repair on semen analysis. They pooled 22 studies of various designs, including meta-analyses as well as randomized and nonrandomized prospective controlled studies, and analyzed sperm concentration before and after repair of clinical varicoceles in men with infertility and abnormal semen parameters. The authors found an overall increase in sperm concentration of 12.32 × 106 ml-1 from before to after interventions. In their study, sperm motility data were available from 17 prospective studies. Using the random-effects model a combined increment of 10.86% in motility was demonstrated. They also evaluated five prospective studies reporting the percentage of progressive motile sperm and confirmed that a significant improvement has occurred as well. The pooled improvement in progressive sperm motility was 9.69% using the random-effects model.

Finally, Schauer et al. published a meta-analysis aiming to determine the impact of each type of intervention; namely, high ligation, inguinal varicocelectomy, and subinguinal varicocelectomy on the semen parameters of subfertile men. The aforementioned study pooled 14 articles including randomized controlled trials, interventional trials, and cohort studies, which accounted for 1476 subjects. Inclusion criteria comprised subfertility and/or at least one abnormal semen parameter, clinical varicocele, and 19 years of age or older. All the studied techniques led to a significant improvement in sperm count and motility. Only minimal differences were observed between intervention groups. The higher increment in sperm count and sperm motility was achieved by inguinal approaches, albeit of no clinical significance when compared to other techniques. The results of this meta-analysis indicated that varicocelectomy leads to significant improvements in sperm count and motility regardless of the chosen surgical technique.

Impaired venous drainage causes an increase in venous stasis and a decrease in arterial blood flow, thus inducing hypoxia, deficiency in testicular microcirculation and subsequent accumulation of oxygen free radicals.

ELIGIBILITY:
Inclusion Criteria:

• Patients with subfertility in different age groups with either unilateral or bilateral clinical varicoceles and at least one abnormal semen parameter.

Exclusion Criteria:

* Patients with varicocele with normal semen parameters.
* Fertile Patients with varicoceles seeking operation only to relieve pain and heaviness.
* Patients with recurrent varicoceles after operation.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian Population , Random Selection of 50 patients with varicocele in the waiting list of varicocelectomy either open or laparoscopic approaches
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate testicular perfusion before and after varicocelectomy | baseline
  Evaluation of testicular perfusion is done by Comparison between Doppler sonographic Parameters Peak systolic velocity ( Cm / sec) , End diastolic velocity ( Cm / sec) , Pulsatility index , And Resistive index Values Before and after varicocelectomy Operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine of Assuit, Asyut, Egypt

REFERENCES:
- [Background] Tarhan S, Ucer O, Sahin MO, Gumus B. Long-term effect of microsurgical inguinal varicocelectomy on testicular blood flow. J Androl. 2011 Jan-Feb;32(1):33-9. doi: 10.2164/jandrol.109.009977. Epub 2010 Jul 29. PMID 20671143
- [Background] Zhang M, Du L, Liu Z, Qi H, Chu Q. The effects of varicocelectomy on testicular arterial blood flow: laparoscopic surgery versus microsurgery. Urol J. 2014 Nov 1;11(5):1900-6. PMID 25361712
- [Background] Akand M, Koplay M, Islamoglu N, Altintas E, Kilic O, Gul M, Kulaksizoglu H, Sivri M, Goktas S. Color Doppler ultrasound characteristics after subinguinal microscopic varicocelectomy. Med Ultrason. 2017 Jan 31;19(1):59-65. doi: 10.11152/mu-920. PMID 28180198